CLINICAL TRIAL: NCT06117111
Title: The Use of Portable Wireless Monitor in Patient Vital Sign Monitoring
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: PAMO2023
Record Dates: First submitted 2023-05-05; First posted 2023-11-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Vital Signs
Keywords: vital signs; intraoperative monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Age: minimum of 18 years, Undergoing pancreatic or ENT tumour surgery, Ability to give informed consent, Volunteering to the study. Monitored in addition to standard monitoring using PaMo device.
  Interventions: Device: PaMo monitoring device

INTERVENTIONS:
Device: PaMo monitoring device — Comparison of the device to standard monitoring

SUMMARY:
This clinical investigation assesses the performance of PaMo patient monitor system (PaMo) and its wearable sensing devices that combines continuous IP, ECG and PPG in detecting developing respiratory depression episodes. PaMo patient monitor system consists of a wearable measurement unit worn on a patient, bedside mobile unit that receives the data from the wearable unit through Bluetooth Low Energy connection, visualises it, and can be relayed further to the central unit through WiFi network.

DETAILED DESCRIPTION:
Monitoring of voluntary subjects undergoing major surgery requiring postoperative intensive care treatment with PaMo patient monitoring device that includes continuous ECG, respiration and PPG monitoring.

The monitoring device is connected during anaesthesia preparation before induction of general anaesthesia and monitoring is continued throughout the surgery and in the intensive care unit (ICU) for total of 24 hours. For reference data, GE Carescape B850 patient monitors are used continuously for oxygen saturation, ECG and respiration signals. The data are collected from the reference patient monitor using a S/5 collect software and a study computer. In addition, to obtain a gold standard reference for SpO2 with blood gas analyzer arterial samples are taken every two hours during anesthesia and in the ICU concurrently with the routine checkups. During the surgery, an arterial cannula collects continuous blood pressure data and can be used for taking blood samples. The data collected with PaMo device and reference monitor are analyzed in Tampere University by researchers and used in device, software and algorithm development.

User experience information and usability feedback are collected at the end of the study from the medical staff with an interview form.

The study does not include a control group. All subjects are using the devices in similar way and the parameters collected from the same individual using two different methods are compared.

ELIGIBILITY:
Inclusion Criteria:

* Age: minimum of 18 years
* Undergoing pancreatic or ENT tumour surgery
* Ability to give informed consent
* Volunteering to the study

Exclusion Criteria:

* Age under 18 years
* Insufficient knowledge in Finnish
* Cardiac pacemaker
* Inability to give informed consent
* Denial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The main study population is formed by adult patients entering to pancreatic or ear tumour surgery following postoperative intensive care treatment.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Electrocardiography (ECG) | Continuous measurement 24 hours
  Mean error an mean absolute error between the study device and standard monitor heart rae
Plethysmography | Continuous measurement 24 hours
  Mean error and mean absolute error between the study monitor and standard monitor
Respiration rate | Continuous measurement 24 hours
  Mean error and mean absolute error between the study monitor and standard monitor

SECONDARY OUTCOMES:
usability | Continuous measurement 24 hours
  usability of the evaluated patient monitoring solution for showing its usability, understandable user interface, suitability of the materials, unobtrusiveness, and fulfilment of related design input requirements. Questionnaire results
blood pressure | Continuous measurement 24 hours
  blood pressure Mean error and mean absolute error between the study monitor and standard monitor and algorithm development

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Harju, Principal Investigator — Deputy chief physician
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No